CLINICAL TRIAL: NCT06596642
Title: Taiwan β-Thalassemia Major Real-World Study for Luspatercept
Brief Title: A Real-World Study of β-Thalassemia Major Treatment With Luspatercept in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA056-1132
Record Dates: First submitted 2024-07-29; First posted 2024-09-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: β-Thalassemia Major
Keywords: β-Thalassemia major
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Adults participants diagnosed with β-thalassemia major
  Interventions: Drug: Luspatercept

INTERVENTIONS:
Drug: Luspatercept — As per product label

SUMMARY:
This real-world study will assess the efficacy and safety of luspatercept treatment for β-thalassemia major in Taiwan as well as the impact on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age.
* Participants with the diagnosis of transfusion-dependent β-thalassemia major who are eligible to the treatment of luspatercept.
* Before luspatercept treatment, participant's transfusion burden ≥ 24 Red Blood Cell units in 24 weeks, without ≥35-day transfusion free.

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients.
* Pregnancy.
* Participants requiring treatment to control the growth of extramedullary hematopoiesis (EMH) masses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults participants in Taiwan diagnosed with β-thalassemia major and treated with luspatercept.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Number of Red Blood Cell (RBC) transfusion units received by participants | Baseline, every 3 weeks thereafter until week 96
Participant hemoglobin (Hb) level results | Baseline, every 3 weeks thereafter until week 96
Participant serum ferritin results | Baseline, week 12, 24, 36, 48, 60, 72, 84 and 96

SECONDARY OUTCOMES:
Participant platelet level results | Baseline, and every 3 weeks thereafter up to week 96
Participant white blood cell count results | Baseline, and every 3 weeks thereafter up to week 96
Participant reticulocytes/normoblast count results | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Participant Hemoglobin F (HbF) levels | Baseline and weeks 6 and 12
Participant uric acid level results | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Participant lactate dehydrogenase (LDH) level results | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Participant aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ratio | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Participant creatinine level results | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Participant bilirubin (total and direct) laboratory values | Baseline, and weeks 12, 24, 36, 48, 60, 72, 84 and 96
Type of iron chelating therapy prescribed to participants | Baseline, every 3 weeks thereafter until week 96
Iron chelating therapy treatment dosage prescribed to participants | Baseline, every 3 weeks thereafter until week 96
Participant Adverse Events (AEs) | Baseline and every 3 weeks until week 12, then weeks 24, 36, 48, 60, 72, 84 and 96
Participant health-related quality of life as assessed by Transfusion-dependent Quality of Life (TranQoL) questionnaire | Baseline, week 12, 24, 48, 72 and 96
Participant health-related quality of life as assessed by EQ-5D-5L questionnaire | Baseline, week 12, 24, 48, 72 and 96
Luspatercept treatment dosage prescribed to participants | Baseline, every 3 weeks thereafter until week 96
Duration of luspatercept treatment | Baseline, every 3 weeks thereafter until week 96
Participant reason(s) for luspatercept treatment discontinuation as assessed by the treating clinician | Baseline, every 3 weeks thereafter until week 96
Participant demographics | Baseline
Participant weight | Baseline
Participant β0/β0 genotype status | Baseline
Participant disease status | Baseline
Participant comorbidities | Baseline
Participant concomitant medication | Baseline
Participant β-thalassemia treatment history | Baseline
Participant surgical history (splenectomy and/or cholecystectomy) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- Taiwan (5):
  - Local Institution - 02, Kaohsiung City
  - Local Institution - 04, Tainan
  - Local Institution - 01, Taipei
  - Local Institution - 03, Taipei
  - Local Institution - 05, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/safety/recalls-market-withdrawals-safety-alerts